CLINICAL TRIAL: NCT06624826
Title: Difference in Visual Performance of a Refractive Extended Depth of Focus Intraocular Lens in an Emmetropic or Monovision Modality
Brief Title: Visual Performance of an Extended Depth of Focus IOL in an Emmetropic or Monovision Modality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PureSee MiniMonovision
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PureSee Emmetropia (Experimental): Patient will receive the PureSee IOL with an emmetropic modality
  Interventions: Device: Emmetropic modality
- PureSee Monovision (Experimental): Patient will receive the PureSee IOL in a monovision modality
  Interventions: Device: Monovision modality

INTERVENTIONS:
Device: Emmetropic modality — PureSee IOL, emmetropic modality
  Arms: PureSee Emmetropia
Device: Monovision modality — PureSee IOL, monovision modality
  Arms: PureSee Monovision

SUMMARY:
Comparison of the visual performance of a refractive extended depth of focus intraocular lens in an emmetropic or monovision modality

DETAILED DESCRIPTION:
With an expanding market of different types of intraocular lenses (IOL), spectacle independence is a rising aim in modern cataract surgery. The procedure has in many cases changed from a vision restoring to a presbyopia correcting approach. Although bilateral monofocal IOL implantation, aiming for emmetropia, leads to high levels of patient satisfaction for distance vision, spectacle dependence for reading and intermediate vision tasks is the usual result.

The option commonly used to achieve spectacle independence at intermediate distance (e.g., PC work) is the implantation of enhanced depth of focus (EDOF) IOLs. These IOLs have an extended far focus area which reaches to the intermediate distance, providing high-quality vision over a continuous range of focus, rather than distinct foci with blur in between. In the last years several technologies for EDOF IOLs appeared on the market. The spectrum ranges from small aperture design, bioanalogic design, to diffractive and non-diffractive optics. The disadvantage compared to monofocal lenses in all the technologies mentioned is the potentially worse distance vision and contrast sensitivity as well as dysphotopsia.

A new refractive EDOF lens segment with an extended depth of vision was introduced which promises an increased range of functional vision and less dysphotopsias compared to diffractive EDOF lenses. These non-diffractive IOLs are believed to be a presbyopia correcting alternative for people with existing corneal or macula pathologies, which would preclude them from receiving premium lenses because of the loss of light in the diffractive process. To increase spectacle independence for these patients, IOLs may be used in a monovision modality, with an offset of up to 1.5dpt. This method showed good results in the literature so far for monofocal and multifocal intraocular lenses.

Aim of the study is to compare a new non-diffractive EDOF-IOL, namely the PureSee, set for emmetropia or monovision.

120 eyes of 60 patients will be included into this study. Patients will be either randomized in the emmetropia or the monovision group

Follow-up visits will be 1 week after each surgery and 3 months post-surgically. During these visits, the clinical variables to be assessed will be visual acuity, stereopsis, contrast sensitivity, and binocular defocus curves.

ELIGIBILITY:
Inclusion Criteria:

* Age-related bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* Axial length: 21.00-27.00mm
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically relevant
* Written informed consent prior to surgery

Exclusion Criteria:

* Active ocular disease (e.g chronic uveitis, diabetic retinopathy, chronic glaucoma not responsive to medication, corneal dystrophies, etc.) precluding good post-operative visual acuity
* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX)
* Irregular astigmatism on corneal tomography
* Pronounced dry eye disease
* Previous ocular surgery or trauma
* Persons who are pregnant or nursing (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Corrected and uncorrected binocular visual acuity for near distance | 12 months
  Corrected and uncorrected binocular visual acuity for near distance will be assessed at 40 cm using ETDRS charts

SECONDARY OUTCOMES:
Corrected and uncorrected binocular visual acuity for distance | 12 months
  Corrected and uncorrected binocular visual acuity for distance will be assessed at 4 m using ETDRS charts
Corrected and uncorrected binocular visual acuity for intermediate distance | 12 months
  Corrected and uncorrected binocular visual acuity for intermediate distance will be assessed at 66 cm using ETDRS charts
Contrast sensitivity | 12 months
  Contrast sensitivity will be tested using the Optec Vision tester under mesopic and photopic conditions with and without an additional glare source
Subjective quality of vision | 12 months
  Subjective quality of vision will be assessed using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery (VIROS)
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided